CLINICAL TRIAL: NCT03444870
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Efficacy, and Safety Study of Gantenerumab in Patients With Early (Prodromal to Mild) Alzheimer's Disease
Brief Title: Efficacy and Safety Study of Gantenerumab in Participants With Early Alzheimer's Disease (AD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision to terminate development of Gantenerumab for treatment of prodromal/mild/early-stage Alzheimer's disease following results of a pre-planned analysis of the safety and efficacy of Gant in Graduate I&II (WN29922/WN39658).
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN29922; 2017-001364-38 (EudraCT Number)
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — gantenerumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gantenerumab (Experimental): Gantenerumab will be administered as SC injections with gradual uptitration.
  Interventions: Drug: Gantenerumab
- Placebo (Placebo Comparator): Placebo will be administered as SC injections with gradual uptitration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gantenerumab — Gantenerumab will be administered as per the schedule specified in the respective arm.
  Other Names: RO4909832
  Arms: Gantenerumab
Drug: Placebo — Placebo will be administered as per the schedule specified in the respective arm.
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel-group study will evaluate the efficacy and safety of gantenerumab versus placebo in participants with early (prodromal to mild) AD. All participants must show evidence of beta-amyloid pathology. Eligible participants will be randomized 1:1 to receive either subcutaneous (SC) injection of gantenerumab or placebo. The primary efficacy assessment will be performed at the end of the double blind period at week 116. Participants will then be offered to enter into an open-label extension (OLE). Participants not willing to go to the OLE will participate in a long term follow-up period for up to 50 weeks after the last gantenerumab dose.

ELIGIBILITY:
Key Inclusion criteria:

* Meets National Institute on Aging/Alzheimer's Association (NIAAA) core clinical criteria for probable AD dementia or prodromal AD (consistent with the NIAAA diagnostic criteria and guidelines for mild cognitive impairment)
* Evidence of the AD pathological process, as confirmed by CSF tau/A-beta42or amyloid PET scan
* Demonstrated abnormal memory function
* MMSE score greater than or equal to 22 (≥ 22)
* Clinical dementia rating-global score (CDR-GS) of 0.5 or 1.0
* Availability of a reliable study partner who accepts to participate in study procedures throughout the 2 years duration of study
* If receiving symptomatic AD medications, the dosing regimen must have been stable for 3 months prior to screening and until randomization
* For enrollment in the China extension, patients must have residence in mainland China, Hong Kong, or Taiwan and be of Chinese ancestry
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods

Key Exclusion criteria:

* Any evidence of a condition other than AD that may affect cognition
* History of schizophrenia, schizoaffective disorder, major depression, or bipolar disorder
* History or presence of clinically evident systemic vascular disease that in the opinion of the investigator has the potential to affect cognitive function
* History or presence of clinically evident cerebrovascular disease
* History or presence of posterior reversible encephalopathy syndrome
* History or presence of any stroke with clinical symptoms within the past 12 months, or documented history within the last 6 months of an acute event that is consistent with a transient ischemic attack
* History of severe, clinically significant CNS trauma
* History or presence of intracranial mass (e.g., glioma, meningioma) that could potentially impair cognition
* Presence of infections that affect brain function or history of infections that resulted in neurologic sequelae
* History or presence of systemic autoimmune disorders that potentially cause progressive neurologic disease with associated cognitive deficits
* At risk for suicide in the opinion of the investigator
* Alcohol and/or substance abuse or dependants in past 2 years
* Relevant brain hemorrhage, bleeding disorder and cerebrovascular abnormalities
* Any contraindications to brain MRI
* Unstable or clinically significant cardiovascular, kidney or liver disease
* Uncontrolled hypertension
* Unstable or clinically significant cardiovascular disease
* Abnormal thyroid function
* Patients with evidence of folic acid deficiency

Exclusion for Open-Label Extension (OLE):

* Discontinued from study treatment during the double-blind treatment period
* Received any other investigational medication during the double-blind treatment period or after the end of double-blind treatment
* Participation in the OLE deemed inappropriate by the investigator
* Presence of ARIA-E findings at the Week 116 MRI scan

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (172):
- United States (33):
  - Center for Neurosciences, Tucson, Arizona
  - Global Clinical Trials; Irvine, CA, Irvine, California
  - Sutter Medical Group, Neurology, Sacramento, California
  - Syrentis Clinical Research, Santa Ana, California
  - California Neuroscience Research Medical Group, Inc, Sherman Oaks, California
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - JEM Research LLC, Atlantis, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Alzheimer?s Research and Treatment Center, Wellington, Florida
  - Columbus Memory Center, Columbus, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Southern Illinois University, School of Medicine, Springfield, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Via Christi Research, Wichita, Kansas
  - Precise Research Centers, Flowood, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Neurological Associates of Long Island, PC, Lake Success, New York
  - Columbia University Medical Center, New York, New York
  - Ohio State University; College of Medicine, Columbus, Ohio
  - Abington Neurological Associates, Abington, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Drexel University; College of Medicine, Philadelphia, Pennsylvania
  - Coastal Neurology, Port Royal, South Carolina
  - Senior Adults Specialty Research, Austin, Texas
  - Neurology Consultants of Dallas; Research Department, Dallas, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Neurology Specialists, Norfolk, Virginia
  - Neurological Associates, Inc., Richmond, Virginia
  - National Clinical Research Inc.-Richmond, Richmond, Virginia
  - UW Wisconsin-Madison, Madison, Wisconsin
- Australia (7):
  - St Vincent's Hospital Sydney; Neurology, Darlinghurst, New South Wales
  - Central Coast Neurosciences Research, Erina, New South Wales
  - Southern Neurology, Kogarah, New South Wales
  - The Queen Elizabeth Hospital; Neurology, Woodville, South Australia
  - Heidelberg Repatriation Hospital; Medical and Cognitive Research Centre, Heidelberg West, Victoria
  - Neuro Trials Victoria, Noble Park, Victoria
  - Australian Alzheimer's Research Foundation, Nedlands, Western Australia
- Brazil (6):
  - Hospital Nossa Senhora das Graças; Setor de Pesquisa em Neurologia, Curitiba, Paraná
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Clinica Clinilive ltda, Maringá, Paraná
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Clínica Dr. Norton Sayeg LTDA - EPP, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP_X; Neurologia, São Paulo, São Paulo
- Canada (11):
  - Medical Arts Health Research Group, Penticton, British Columbia
  - The Medical Arts Health Research Group - West Vancouver, Vancouver, British Columbia
  - Parkwood Hospital; Geriatric Medicine, London, Ontario
  - Centre for Memory and Aging, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael'S Hospital, Toronto, Ontario
  - Baycrest Health Sciences, Toronto, Ontario
  - Devonshire Clinical Research, Woodstock, Ontario
  - Center for Diagnosis and Research on Alzheimer's disease, Greenfield Park, Quebec
  - Q & T Research Sherbrooke, Sherbrooke, Quebec
  - Alpha Recherche Clinique, Québec
- China (28):
  - China-Japan Friendship Hospital, Beijing
  - Beijing Anding Hospital, Capital Medical University, Beijing
  - Beijing Tian Tan Hospital,Capital Medical University, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - Sun Yat-sen Memorial Hospital; Neurology, Guangzhou
  - Guangdong Provincial People's Hospital; Breast, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - The Second Affiliated Hospital, Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Zhongda Hospital Affiliated to Southeast University, Nanjing
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Mental Health Center, Shanghai
  - Huashan Hospital Affiliated to Fudan University, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Sixth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - The University of Hong Kong-Shenzhen Hospital; Local Ethic Committee, Shenzhen
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical College, Wenzhou
  - Northern Jangsu People's Hospital, Yangzhou
  - Henan Provincial People's Hospital, Zhengzhou
- France (9):
  - CHU Amiens Hopital Sud; Neurologie, Amiens Cedex1
  - Hôpital Avicenne; Centre de Recherche Clinique, Bobigny
  - Groupement Hospitalier Est - Hôpital Neurologique; Neurologie A (U502), Bron
  - CHU de la Timone - Hopital d Adultes; Service de Neurologie, Marseille
  - Hôpital Lariboisière, Paris
  - CHU Poitiers - Hopital La Miletrie, Poitiers
  - CHU Strasbourg Hôpital Hautepierre, Strasbourg
  - Gerontopole; Centre de Recherche clinique, Toulouse
  - Hopital des Charpennes, Villeurbanne
- Germany (12):
  - Ambulates Gesundheitszentrum der Charité GmbH; MVZ Neurologie Campus Benjamin Franklin, Berlin
  - ECRC Experimental and Clinical Research Center, Charité Campus Berlin Buch, Memory Clinic, Berlin
  - St. Josef-Hospital, Klinik für Neurologie, Bochum
  - Universitätsklinikum Köln; Klinik und Poliklinik für Psychiatrie und Psychotherapie, Cologne
  - PANAKEIA - Arzneimittelforschung Leipzig GmbH, Leipzig
  - Universitätsmedizin derJohannes Gutenberg-Universität Mainz;Klinik für Psychiatrie und Psychotherapi, Mainz
  - Klinikum rechts der Isar der TU München; Klinik für Psychiatrie und Psychotherapie, München
  - Universitätsklinikum Münster; Klinik und Poliklinik für Neurologie, Münster
  - Universitätsklinikum Rostock Zentrum für Nervenheilkunde, Rostock
  - Universitätsklinikum Ulm; Klinik für Neurologie, Ulm
  - Studienzentrum Nordwest Dr med Joachim Springub Herr Wolfgang Schwarz, Westerstede
  - Forschungszentrum Ruhr, Witten
- Semmelweis University; Department of Neurology, Budapest, Hungary
- Italy (10):
  - Nuovo Ospedale Civile S. Agostino-Estense; Clinica Neurologica ? Dipartimento di Neuroscienze, Modena, Emilia-Romagna
  - Fondazione Santa Lucia IRCCS; Neurologia e Riabilitazione Neurologica, Rome, Lazio
  - Umberto I Policlinico di Roma-Università di Roma La Sapienza, Rome, Lazio
  - Ospedale San Giovanni Calibita Fatebenefratell;Neurologia, Rome, Lazio
  - IRCCS ?Centro S. Giovanni di Dio? Fatebenefratelli -UO Alzheimer, Brescia, Lombardy
  - IRCCS Ospedale San Raffaele; Centro Disturbi della Memoria, Milan, Lombardy
  - ASST DI MONZA; Neurologia, Monza, Lombardy
  - IRCCS Neuromed; Neurologia I-Centro studio e cura delle demenze e UVA, Pozzilli, Molise
  - AO Città della Salute e della Scienza Osp.S.Giov.Battista Molinette; SC Geriatria, Turin, Piedmont
  - Dipartimento delle Patologie Emergenti; Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo, Sicily
- Japan (18):
  - Medical Corporation Hakuyokai Kashiwado Hospital, Chiba
  - Inage Neurology and Memory Clinic, Chiba
  - Juntendo University Urayasu Hospital, Chiba
  - Southern Tohoku Medical Clinic, Fukushima
  - Yuai Clinic, Kanagawa
  - Shonan Kamakura General Hospital, Kanagawa
  - Mishima Hospital, Niigata
  - NHO Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka
  - Shizuoka City Shimizu Hospital, Shizuoka
  - Jichiidai Station Brain Clinic, Tochigi
  - Yotsuya Medical Cube, Tokyo
  - Tokyo Medical and Dental University Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Tokyo Metropolitan Geriatric Hospital, Tokyo
  - Nozomi Memory Clinic, Tokyo
  - National Center of Neurology and Psychiatry, Tokyo
  - P-One Clinic, Tokyo
  - Yamagata Tokusyukai Hospital, Yamagata
- Vilnius University Hospital Santariskiu Clinics; Neurology, Vilnius, Lithuania
- Peru (4):
  - Hospital IV Alberto Sabogal Sologuren; Unidad de Investigacion, Bellavista
  - Clinica Internacional; Unidad De Investigacion, Lima
  - Hospital Nacional Dos de Mayo; Unidad de Investigacion de Neurologia, Lima
  - Hospital Nacional Cayetano Heredia; Servicio de Neurologia, San Martín de Porres
- Russia (9):
  - FSBHI Siberian Clinical Center of the Federal Medical and Biological Agency, Krasnoyarsk, Krasnoyarsk Krai
  - University ?linic of headaches, Moscow, Moscow Oblast
  - City Clin Hosp n.a. S.P.Botkin, Moscow, Moscow Oblast
  - Central Clinical Hospital #2 N.A. Semashko OAO RJHD, Moskva, Moscow Oblast
  - Russian Medical Military Academy n.a. S.M.Kirov; Neurology Department, Saint Petersburg, Sankt-Peterburg
  - Vertebronevrologiya LLC, Kazan', Tatarstan Republic
  - State autonomous institution of healthcare Inter-regional clinical and diagnostic center, Kazan', Tatarstan Republic
  - City Clinical Hospital # 2 n.a. V.I. Razumovsky, Saratov
  - Nebbiolo Center for Clinical Trials, Tomsk
- Spain (17):
  - Hospital Universitari de Bellvitge; Servicio de Neurologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital General De Catalunya; Servicio de Neurologia, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario Marques de Valdecilla; Servicio de Neurología, Santander, Cantabria
  - Hospital San Pedro; Servicio de Neurología, Logroño, La Rioja
  - HM Universitario Puerta del Sur CINAC (C.Integ.Neuroc);; Servicio de Psiquiatría, Móstoles, Madrid
  - Hospital General Universitario de Albacete; Servicio de Neurología, Albacete
  - Hospital Vall d'Hebron; Servicio de Neurología, Barcelona
  - Hospital Clinic i Provincial; Servicio de Neurologia, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Neurologia, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Neurologia, Córdoba
  - Hospital Ramon y Cajal; Servicio de Neurologia, Madrid
  - Hospital Ruber Internacional; Servicio de Neurología, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Neurologia, Madrid
  - Complejo Asistencial Universitario de Salamanca; Servicio de Psiquiatría, Salamanca
  - Hospital Virgen del Rocío; Servicio de Neurología, Seville
  - Hospital Universitario Dr. Peset; Servicio de Neurologia, Valencia
  - Servicio de Neurología Hospital Viamed Montecanal., Zaragoza
- Taiwan (6):
  - Changhua Christian Hospital; Neurology, Changhua County
  - Kaohsiung Medical University Hospital; Neurology, Kaohsiung City
  - Chang Gung Memorial Foundation - Kaohsiung - Neurology, Niaosong Dist.
  - China Medical University Hospital; Neurology, North Dist.
  - National Taiwan University Hospital; Neurology, Taipei
  - Chang Gung Memorial Foundation - Linkou - Neurology, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Chandler JM, Lansdall CJ, Ye W, McDougall F, Belger M, Toth B, Mi X, Sink KM, Atkins AS. The Alzheimer's Disease Cooperative Study - Activities of Daily Living dependence score: revision and validation of an algorithm evaluating patient dependence across the spectrum of AD severity. J Prev Alzheimers Dis. 2025 Sep;12(8):100261. doi: 10.1016/j.tjpad.2025.100261. Epub 2025 Jul 1. PMID 40603145
- [Derived] Asada T, Thanasopoulou A, Delmar P, Wojtowicz J, Smith J, Yoshiyama Y, Yokoi K, Watanabe C, Isozaki M, Ozaki R, Ishida T, Tatsuda H, Tamaoka A. Japanese participant data from three gantenerumab trials in early Alzheimer's disease. Alzheimers Dement. 2025 Apr;21(4):e70192. doi: 10.1002/alz.70192. PMID 40302041
- [Derived] Bittner T, Tonietto M, Klein G, Belusov A, Illiano V, Voyle N, Delmar P, Scelsi MA, Gobbi S, Silvestri E, Barakovic M, Napolitano A, Galli C, Abaei M, Blennow K, Barkhof F. Biomarker treatment effects in two phase 3 trials of gantenerumab. Alzheimers Dement. 2025 Feb;21(2):e14414. doi: 10.1002/alz.14414. Epub 2025 Jan 30. PMID 39887500
- [Derived] Salloway S, Wojtowicz J, Voyle N, Lane CA, Klein G, Lyons M, Rossomanno S, Mazzo F, Bullain S, Barkhof F, Bittner T, Schneider A, Grundman M, Aldea R, Boada M, Smith J, Doody R. Amyloid-Related Imaging Abnormalities (ARIA) in Clinical Trials of Gantenerumab in Early Alzheimer Disease. JAMA Neurol. 2025 Jan 1;82(1):19-29. doi: 10.1001/jamaneurol.2024.3937. PMID 39556389
- [Derived] Bateman RJ, Smith J, Donohue MC, Delmar P, Abbas R, Salloway S, Wojtowicz J, Blennow K, Bittner T, Black SE, Klein G, Boada M, Grimmer T, Tamaoka A, Perry RJ, Turner RS, Watson D, Woodward M, Thanasopoulou A, Lane C, Baudler M, Fox NC, Cummings JL, Fontoura P, Doody RS; GRADUATE I and II Investigators and the Gantenerumab Study Group. Two Phase 3 Trials of Gantenerumab in Early Alzheimer's Disease. N Engl J Med. 2023 Nov 16;389(20):1862-1876. doi: 10.1056/NEJMoa2304430. PMID 37966285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study at 137 sites across 15 countries (Australia, Brazil, Canada, China, France, Germany, Hungary, Italy, Japan, Lithuania, Peru, Russia, Taiwan, Spain, and the United States) during the global phase. Participants were enrolled at 21 sites in China during the China extension phase of the study.
  The open-label period in China was not started as the study was terminated early by the Sponsor.
Pre-assignment Details: A total of 985 participants with early (prodromal to mild) Alzheimer's Disease (AD) were randomized to either the gantenerumab (n=499) or placebo arm (n=486) to enter the double-blind treatment (DBT) period of the global phase. A total of 68 early (prodromal to mild) AD participants were randomized to the gantenerumab (n=35) or placebo arm (n=33) to enter the DBT period of the China extension phase.
Groups:
- Global - DBT Period: Placebo: Participants received gantenerumab matching placebo, SC injection, every four weeks (Q4W) up to Week 36 and then every two weeks (Q2W) up to approximately 114 weeks of the DBT period.
- Global - DBT Period: Gantenerumab: Participants received gantenerumab, SC injection with gradual up-titration starting at a dose of 120 milligrams (mg), Q4W for 3 doses, followed by 255 mg, Q4W for 3 doses, and 510 mg, Q4W for 3 doses, and 510 mg, Q4W for 3 doses. Following this, from Week 36 onwards, participants received gantenerumab, SC injection at a dose of 510 mg, Q2W up to Week 114 of the DBT period.
- China Extension - DBT Period: Placebo: Participants received gantenerumab matching placebo, SC injection, Q4W up to Week 36 and then Q2W up to approximately 110 weeks of the DBT period.
- China Extension - DBT Period: Gantenerumab: Participants received gantenerumab, SC injection with gradual up-titration starting at a dose of 120 mg, Q4W for 3 doses, followed by 255 mg, Q4W for 3 doses, and 510 mg, Q4W for 3 doses. Following this, from Week 36 onwards, participants received gantenerumab, SC injection at a dose of 510 mg, Q2W up to approximately 110 weeks of the DBT period.
- Global - OLE Period: Placebo (DBT) to Gantenerumab: Participants who received gantenerumab matching placebo in the DBT period received gantenerumab SC injections with gradual up titration starting at a dose of 120 mg, Q4W for 3 doses, followed by 255 mg, Q4W for 3 doses, and then at a dose of 510 mg, Q4W up to Week 34 of the OLE period. To maintain the blind to previous treatment assignment, participants received Q2W, SC injections, with alternate doses containing gantenerumab matching placebo.
- Global - OLE Period: Gantenerumab (DBT) to Gantenerumab: Participants who received gantenerumab in the DBT period continued receiving gantenerumab, SC injections, 510 mg, Q2W up to Week 34 of the OLE period.
Period: Double-Blind Treatment (DBT) Period
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab | Global - OLE Period: Placebo (DBT) to Gantenerumab | Global - OLE Period: Gantenerumab (DBT) to Gantenerumab
Started | 486 | 499 | 33 | 35 | 0 | 0
Intent-to-treat (ITT) Analysis Set (ITT analysis set included all participants randomized during the global phase, who received at least one dose of study drug.) | 485 | 499 | 0 | 0 | 0 | 0
Safety-evaluable (SE) Analysis Set (SE analysis set included all participants randomized during the global phase who received at least one dose of study drug. In the DBT period, 4 participants randomized to placebo arm received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety evaluable set, of which 1 participant entered OLE period.) | 481 | 503 | 0 | 0 | 0 | 0
ITT Analysis Set (China) (ITT analysis set (China) included all participants enrolled in China in the China extension phase who received at least one dose of study drug.) | 0 | 0 | 33 | 35 | 0 | 0
SE Analysis Set (China) (SE analysis set (China) included all participants enrolled in China in the China extension phase who received at least one dose of study drug.) | 0 | 0 | 33 | 35 | 0 | 0
Safety Magnetic Resonance Imaging (MRI)-Evaluable (SEMRI) Analysis Set (SEMRI analysis set included all participants in the SE analysis set who had at least one post-baseline safety MRI scan.) | 476 | 497 | 0 | 0 | 0 | 0
Completed | 387 | 375 | 0 | 0 | 0 | 0
Not Completed | 99 | 124 | 33 | 35 | 0 | 0
Not completed — Study Terminated By Sponsor | 0 | 0 | 30 | 35 | 0 | 0
Not completed — Reason not Specified | 17 | 16 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 56 | 63 | 2 | 0 | 0 | 0
Not completed — Protocol Deviation | 4 | 3 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 11 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 10 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 29 | 0 | 0 | 0 | 0
Not completed — Randomized, but not Treated | 1 | 0 | 0 | 0 | 0 | 0
Period: Open-Label Extension (OLE) Period
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab | Global - OLE Period: Placebo (DBT) to Gantenerumab | Global - OLE Period: Gantenerumab (DBT) to Gantenerumab
Started | 0 (Participants who completed the DBT Period were given the option to enroll in the OLE Period to receive gantenerumab.) | 0 (Participants who completed the DBT Period were given the option to enroll in the OLE Period to receive gantenerumab.) | 0 (Participants who completed the China Extension -DBT Period were given the option to enroll in the OLE Period to receive gantenerumab.) | 0 (Participants who completed the China Extension -DBT Period were given the option to enroll in the OLE Period to receive gantenerumab.) | 10 (10 participants who completed the DBT Period enrolled into the OLE Period.) | 19 (19 Participants who completed the DBT Period enrolled into the OLE Period.)
SE Analysis Set (SE analysis set included all participants randomized during the global phase who received at least one dose of study drug. In the DBT period, 4 participants randomized to placebo arm received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety evaluable set, of which 1 participant entered OLE period.) | 0 | 0 | 0 | 0 | 9 | 20
Completed | 0 | 0 | 0 | 0 | 7 | 17
Not Completed | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT analysis set included all participants randomized during the global phase, who received at least one dose of study drug. ITT analysis set (China) included all participants enrolled in China in the China extension phase who received at least one dose of study drug.
Groups:
- Global - DBT Period: Placebo: Participants received gantenerumab matching placebo, SC injection, Q4W up to Week 36 and then Q2W up to approximately 114 weeks of the DBT period.
- Global - DBT Period: Gantenerumab: Participants received gantenerumab, SC injection with gradual up-titration starting at a dose of 120 mg, Q4W for 3 doses, followed by 255 mg, Q4W for 3 doses, and 510 mg, Q4W for 3 doses, and 510 mg, Q4W for 3 doses. Following this, from Week 36 onwards, participants received gantenerumab, SC injection at a dose of 510 mg, Q2W up to Week 114 of the DBT period.
- Total: Total of all reporting groups
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab | Total
Number analyzed (Participants) | 485 | 499 | 33 | 35 | 1052
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (7.8) | 71.1 (7.9) | 65.9 (8.5) | 68.5 (7.3) | 71.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 255 | 290 | 16 | 18 | 579
  Male | 230 | 209 | 17 | 17 | 473
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58 | 52 | 0 | 0 | 110
  Not Hispanic or Latino | 422 | 439 | 32 | 34 | 927
  Unknown or Not Reported | 5 | 8 | 1 | 1 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 18 | 0 | 0 | 36
  Asian | 53 | 52 | 33 | 35 | 173
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 1 | 0 | 0 | 7
  White | 398 | 414 | 0 | 0 | 812
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 14 | 0 | 0 | 24
China Extension: Clinical Dementia Rating-Sum of Boxes (CDR-SB) [Mean (Standard Deviation); unit: score on a scale] — CDR was derived through semi-structured interview with participant and appropriate informant. It rated impairment across 6 domains: memory,orientation,judgment,and problem solving,community affairs,home and hobbies, and personal care on a 5-point scale for which 0=no impairment, 0.5=questionable impairment, and 1, 2, and 3=mild, moderate, severe impairment respectively. The CDR-SB is based on summing each of the domain box scores with total score ranging from 0-18 with higher scores reflecting greater cognitive and functional impairment. Population: ITT analysis set (China) included all participants enrolled in China in the China extension phase who received at least one dose of study drug.
  score on a scale
    number analyzed (Participants) | 0 | 0 | 33 | 35 | 68
    (all) |  |  | 3.29 (1.22) | 3.69 (1.50) | 3.49 (1.38)
DBT Period: CDR-SB [Mean (Standard Deviation); unit: score on a scale] — CDR was derived through semi-structured interview with participant and appropriate informant. It rated impairment across 6 domains: memory,orientation,judgment,and problem solving,community affairs,home and hobbies, and personal care on a 5-point scale for which 0=no impairment, 0.5=questionable impairment, and 1, 2, and 3=mild, moderate, severe impairment respectively. The CDR-SB is based on summing each of the domain box scores with total score ranging from 0-18 with higher scores reflecting greater cognitive and functional impairment. Population: ITT analysis set included all participants randomized during the global phase, who received at least one dose of study drug.
  score on a scale
    number analyzed (Participants) | 485 | 499 | 0 | 0 | 984
    (all) | 3.71 (1.67) | 3.71 (1.57) |  |  | 3.71 (1.62)

OUTCOME MEASURES:

1. Primary Outcome: DBT Period: Change From Baseline to Week 116 in Global Outcome, as Measured by CDR-SB
Description: CDR was derived through semi-structured interview with the participant and an appropriate informant, and it rated impairment across six domains: memory, orientation, judgment, and problem solving, community affairs, home and hobbies, and personal care on a 5-point scale for which 0=no impairment, 0.5=questionable impairment, and 1, 2, and 3=mild, moderate, and severe impairment, respectively. The CDR-SB is based on summing each of the domain box scores with total score ranging from 0-18 with higher scores reflecting greater cognitive and functional impairment. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: ITT analysis set included all participants randomized during the global phase, who received at least one dose of study drug.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 485 | 499
score on a scale | 3.65 (0.16) | 3.35 (0.14)
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; Change from Baseline was calculated based on ANCOVA analysis model which included the following covariates and stratification factors =Treatment + Baseline (BL) + Geographic Region + Disease Stage + AD Medication at BL + Apolipoprotein E, Allele e4 (APOE e4) + Baseline Alzheimer Disease Assessment Scale-Cognition Subscale 13 (ADAS-Cog13) Score + Baseline Alzheimer Disease Cooperative Study Group-Activities of Daily Living (ADCS-ADL); Test type: Superiority; p = 0.0954, ANCOVA; Difference in adjusted mean = -0.31, 95% CI 2-sided [-0.66 to 0.05], Standard Error of Mean 0.18

2. Primary Outcome: China Extension: DBT Period: Change From Baseline to Week 116 in Global Outcome, as Measured by CDR-SB
Description: as for outcome 1
Time Frame: Baseline, Week 116
Population: The study was terminated early by the sponsor before any participant had reached Week 116 visit in the China extension phase.
Arm/Group | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Alzheimer Disease Assessment Scale-Cognition Subscale 13 (ADAS-Cog13) Score
Description: The ADAS-Cog13 total score includes all of the items in the ADAS-Cog11 in addition to delayed word recall and the number cancellation. For the ADAS-cog 13 the range is 0-85 (score range for Delayed Word Recall [DWR] score is 0-10 and for Number Cancellation [NC] is 0-5, thus the score is ADAS-cog 11[0-70] plus the scores for DWR and NC). A higher score indicates worse performance. A negative change from baseline indicates improvement in cognitive function.
Time Frame: Baseline, Week 116
Population: ITT analysis set included all participants randomized during the global phase, who received at least one dose of study drug. Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 480 | 497
score on a scale | 9.82 (0.57) | 8.57 (0.47)
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; Change from BL was calculated based on ANCOVA analysis model which included the following covariates and stratification factors = Treatment + Baseline + Geographical Region + Disease Stage + AD Medication at BL + APOE e4; Test type: Superiority; p = 0.0544, ANCOVA; Difference in adjusted mean = -1.25, 95% CI 2-sided [-2.52 to 0.02], Standard Error of Mean 0.65

4. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Alzheimer's Disease Cooperative Study- Activities of Daily Living (ADCS-ADL) Total Score
Description: ADCS-ADL is a 23-item rater-administered, observer-reported outcome (ObsRO) that captures a participant's ability to perform basic activities of daily living (e.g., eating and toileting) and more complex ADL or instrumental activities of daily living (iADL, e.g., using the telephone, managing finances, preparing a meal). Total score ranges from 0-78, with higher scores reflecting better functioning. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 479 | 497
score on a scale | -12.32 (0.68) | -11.21 (0.60)
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; Change from BL was calculated based on ANCOVA analysis model which included the following covariates and stratification factors = Treatment + Baseline + Region + Disease Stage + AD Medication at BL + APOE e4; Test type: Superiority; p = 0.1729, ANCOVA; Difference in adjusted mean = 1.11, 95% CI 2-sided [-0.48 to 2.70], Standard Error of Mean 0.81

5. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Functional Activities Questionnaire (FAQ) Score
Description: FAQ is a rater-administered ObsRO (informant-based measure) that measures a participant's functional ability to perform complex higher-order activities. The observer provides performance ratings of the target person on ten complex higher-order activities. Total score that ranges from 0-30, with higher scores reflecting greater functional impairment. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 479 | 498
score on a scale | 8.13 (0.33) | 7.28 (0.30)
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0425, ANCOVA; Difference in adjusted mean = -0.86, 95% CI 2-sided [-1.68 to -0.03], Standard Error of Mean 0.42

6. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Mini-Mental State Examination (MMSE) Total Score
Description: MMSE is a rater-administered performance-based outcome (PerfO) that includes a set of standardized questions used to evaluate possible cognitive impairment and help stage the severity level of this impairment. The questions target six areas: orientation, registration, attention, short-term recall, language, and constructional praxis/visuospatial abilities. Total score ranges from 0-30, with lower scores indicating greater impairment. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 485 | 499
score on a scale | -5.18 (0.25) | -4.86 (0.23)
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; Change from Baseline was calculated based on ANCOVA analysis model which included the following covariates and stratification factors =Treatment + Baseline + Geographic Region + Disease Stage + AD Medication at BL + APOE e4; Test type: Superiority; p = 0.2904, ANCOVA; Difference in adjusted mean = 0.32, 95% CI 2-sided [-0.28 to 0.93], Standard Error of Mean 0.31

7. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Alzheimer Disease Assessment Scale-Cognition Subscale 11 (ADAS-Cog11) Score
Description: The ADAS-Cog11 was designed to measure cognitive symptom change in participants with Alzheimer's Disease (AD) and consisted of 11 tasks. The standard 11 items (and corresponding score range) were: word recall (0-10), commands (0-5), constructional praxis (0-5), naming objects and fingers (0-5), ideational praxis (0-5), orientation (0-8), word recognition (0-12), spoken language ability (0-5), comprehension of spoken language (0-5), word-finding difficulty (0-5), and remembering test instructions (0-5). The test included 7 performance items and 4 clinician-rated items. The ADAS-Cog11 total score was the sum of all 11 individual items, with a total score ranging from 0 (no impairment) to 70 (severe impairment). Higher scores indicated more severe cognitive impairment. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 481 | 498
score on a scale | 8.42 (0.52) | 7.44 (0.43)
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.1036, ANCOVA; Difference in adjusted mean = -0.97, 95% CI 2-sided [-2.14 to 0.20], Standard Error of Mean 0.60

8. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Verbal Fluency Task (VFT) Score
Description: VFT is a rater administered PerfO that measures speed and flexibility of verbal thought with a total score that ranges from 0-99 (lower scores indicating lower performance). A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 481 | 499
score on a scale | -3.46 (0.31) | -3.53 (0.30)
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.8468, ANCOVA; Difference in adjusted mean = -0.07, 95% CI 2-sided [-0.79 to 0.65], Standard Error of Mean 0.37

9. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in the Coding (Digit Symbol Substitution Test [DSST]) Subtest
Description: Coding, also called DSST is a rater administered PerfO that measures speed of processing and associative memory with a total score that ranges from 0-135 (lower scores indicating lower performance). The DSST was adapted from the Wechsler Adult Intelligence Scale. The 120-second version of the test was used in this study. Positive change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 480 | 498
score on a scale | -6.47 (0.64) | -6.27 (0.54)
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.8030, ANCOVA; Difference in adjusted mean = 0.20, 95% CI 2-sided [-1.35 to 1.74], Standard Error of Mean 0.79

10. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living (ADCS-iADL) Instrumental Score
Description: The ADCS-iADL measures activities such as using the telephone, shopping and preparing a meal. The ADCS-iADL consists of 16 questions with a score range of 0 to 56 where a higher score represents better function. Positive change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 479 | 497
score on a scale | -10.80 (0.56) | -9.80 (0.51)
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.1439, ANCOVA; Difference in adjusted mean = 1.00, 95% CI 2-sided [-0.34 to 2.34], Standard Error of Mean 0.68

11. Secondary Outcome: DBT Period: Number of Participants With at Least One Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution.
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 131 weeks)
Population: SE analysis set included all participants randomized during the global phase who received at least one dose of study drug. In the DBT period, four participants randomized to placebo arm received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 481 | 503
Participants | 423 | 454

12. Secondary Outcome: DBT Period: Number of Participants With Post-baseline Suicidal Ideation or Suicidal Behavior as Measured Using Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS=assessment tool used to assess lifetime suicidality of a participant (at baseline) as well as any new instances of suicidality (C-SSRS since last visit). Structured interview prompts recollection of suicidal ideation, including intensity of ideation, behavior, & attempts with actual/potential lethality. Categories have binary responses (yes/no) & include Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent, Preparatory Acts and Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. Suicidal ideation/behavior is indicated by a "yes" answer to any of the listed categories. Score of 0 is assigned if no suicide risk is present. Score of 1 or higher= suicidal ideation or behavior. Categories with non-zero values are only reported here.
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 131 weeks)
Population: SE analysis set included all participants randomized during the global phase who received at least one dose of study drug. In the DBT period, four participants randomized to placebo arm received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety analysis set. Overall number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 467 | 489
Participants
  Suicidal Ideation: Passive | 13 | 17
  Suicidal Ideation: Active-Nonspecific | 1 | 3
  Suicidal Ideation: Active-Method, But No Intent or Plan | 6 | 3
  Suicidal Ideation: Active-Method and Intent, But No Plan | 2 | 0
  Suicidal Ideation: Active-Method, Intent, and Plan | 2 | 0
  Suicidal Ideation: No Event | 443 | 466
  Suicidal Behavior: Interrupted Attempt | 0 | 1
  Suicidal Behavior: No Event | 467 | 488
  Self-injurious Behavior Without Suicidal Intent: No Event | 467 | 489

13. Secondary Outcome: DBT Period: Number of Participants With at Least One Amyloid-Related Imaging Abnormalities-Edema (ARIA-E) Magnetic Resonance Imaging (MRI) Finding
Description: ARIA are an identified risk with anti-amyloid antibodies, including gantenerumab. These changes can be identified on brain MRI. In ARIA-E, (E for oedema or effusion), oedema can be seen in different areas of the brain on MRI, representing fluid leakage into the brain parenchyma or sulcal spaces.
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 131 weeks)
Population: SEMRI analysis set included all participants in the SE analysis set who had at least one post-baseline safety MRI scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 476 | 497
Participants | 5 | 105

14. Secondary Outcome: DBT Period: Number of Participants With at Least One Amyloid-Related Imaging Abnormalities-Haemosiderin Deposition (ARIA-H) MRI Finding
Description: ARIA are an identified risk with anti-amyloid antibodies, including gantenerumab. These changes can be identified on brain MRI. ARIA-H (H for hemosiderosis) are small foci of signal loss observed on MRI sequences sensitive for paramagnetic tissue properties and comprise cerebral microbleeds (small foci of bleeding in the brain parenchyma) and leptomeningeal hemosiderosis (small foci of bleeding on the surface of the brain). These changes also occur sporadically in AD.
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 131 weeks)
Population: SEMRI analysis set included all participants in the SE analysis set who had at least one post-baseline safety MRI scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 476 | 497
Participants | 6 | 40

15. Secondary Outcome: DBT Period: Number of Participants With Injection-Site Reactions
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution. Local injection reactions (or injection site reactions) are defined as AEs related to the injection site that occur during or within 24 hours after study drug administration that are judged to be related to the study drug injection.
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 131 weeks)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 481 | 503
Participants | 43 | 94

16. Secondary Outcome: DBT Period: Number of Participants With Anti-Drug Antibodies (ADA) to Gantenerumab
Description: The number of participants with positive results for ADA against gantenerumab at any of the post-baseline assessment time-points were reported. Participant with an ADA assay result from at least one post-baseline sample was defined as a post-baseline evaluable participant. Treatment Emergent ADA = A participant with a negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result.
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 131 weeks)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 489
Participants | 10

17. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Brain Amyloid Load as Measured by Amyloid Positron Emission Tomography (PET) Scan in a Subset of Participants
Description: Brain amyloid load over time was assessed using [18F] florbetaben or [18F] flutemetamol tracers. These are PET radioligand selective to amyloid. Amyloid PET burden was measured in a composite region of interest (ROI) by using standardized uptake value ratio (SUVR) mapped to the centiloid scale. The weighted composite target region are composed of (both left and right side): frontal lobe, parietal lobe, temporal lobe lateral, cingulum posterior and anterior cingulate gyrus. The reference region used to normalize the composite region was the whole cerebellum. The centiloid scale anchor points are 0 and 100, where 0 represents a high-certainty amyloid negative scan and 100 represents the amount of global amyloid deposition found in a typical AD scan.
Time Frame: Baseline, Week 116
Population: Amyloid-PET modified ITT (mITT) analysis set included all participants in the ITT analysis set who participated in the Amyloid-PET substudy and who had at least one Amyloid-PET scan with a valid quantitative measurement performed with either florbetaben or flutemetamol and who did not withdraw from the Amyloid-PET substudy before randomization. Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 41 | 49
score on a scale | 9.06 (3.046) | -57.38 (2.841)
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; Change from BL was calculated based on mixed-effect model of repeated measure which included the following covariates and stratification factors = Baseline + APOE e4 status + Type of Tracer + Analysis Visit + Treatment + Treatment*Analysis Visit + Analysis Visit*Baseline; Test type: Superiority; p < .0001, Mixed Model for Repeated Measures; Difference in adjusted means = -66.44, 95% CI 2-sided [-74.71 to -58.16], Standard Error of Mean 4.171

18. Secondary Outcome: DBT Period: Change From Baseline to Week 116 in Brain Tau Load, as Measured by Tau PET Scan in a Subset of Participants
Description: Change in tau load= how much neurofibrillary tau pathology is present in brain assessed by PET Scan. [18F] GTP1 was the tau PET radioligand. Tau load was measured using SUVR in 4 composite target ROIs: Temporal composite target region (left & right)=anterior & posterior superior temporal gyrus, posterior temporal lobe, fusiform gyrus, & middle & inferior temporal gyrus; Medial temporal composite region excluding hippocampus (left & right): amygdala, parahippocampus & anterior medial & lateral temporal lobe; Frontal lobe (left & right) & Parietal lobe (left & right). Inferior cerebellar grey matter=reference region for calculating SUVRs for all 4 regions. Tau-PET-mITT analysis set=all participants in ITT analysis set who participated in Tau PET sub-study & who had at least one Tau PET scan with a valid quantitative measurement & who did not withdraw from Tau PET substudy before randomization. Overall number analyzed=number of participants with data available for analysis.
Time Frame: Baseline, Week 116
Population: As pre-specified in protocol/SAP, single tau PET substudy analyzed participants from 2 studies i.e. WN29922 (NCT03444870) & WN39658 (NCT03443973), hence data for Tau PET was analyzed at pooled level of WN29922 &WN39658. These studies had identical study design & enrolled an Early AD population. Tau PET analysis was planned in a subset of participants, to get an optimum sample size for analysis, it was pre-planned to conduct 1 tau PET substudy for participants willing to consent to the procedure.
Measure: Mean (Standard Error); unit: SUVR
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 29 | 48
SUVR
  ROI: Temporal Composite Region | 0.12 (0.018) | 0.13 (0.014)
  ROI: Medial Temporal Composite Region [not including the Hippocampus] | 0.08 (0.014) | 0.09 (0.011)
  ROI: Frontal Lobe | 0.08 (0.012) | 0.08 (0.009)
  ROI: Parietal Lobe | 0.09 (0.020) | 0.09 (0.016)
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; Temporal Composite Region: Change from BL was calculated based on mixed-effect model of repeated measure which included the following covariates and stratification factors = Baseline + APOE e4 status + Study + Analysis Visit + Treatment + Treatment*Analysis Visit + Analysis Visit*Baseline; Test type: Superiority; p = 0.7816, Mixed Model for Repeated Measures; Difference in adjusted mean = 0.01, 95% CI 2-sided [-0.04 to 0.05], Standard Error of Mean 0.023
Statistical Analysis 2: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; Medial Temporal Composite Region: Change from BL was calculated based on mixed-effect model of repeated measure which included the following covariates and stratification factors = Baseline + APOE e4 status + Study + Analysis Visit + Treatment + Treatment*Analysis Visit + Analysis Visit*Baseline; Test type: Superiority; p = 0.6203, Mixed Model for Repeated Measures; Difference in adjusted means = 0.01, 95% CI 2-sided [-0.03 to 0.05], Standard Error of Mean 0.018
Statistical Analysis 3: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; Frontal Lobe: Change from BL was calculated based on mixed-effect model of repeated measure which included the following covariates and stratification factors = Baseline + APOE e4 status + Study + Analysis Visit + Treatment + Treatment*Analysis Visit + Analysis Visit*Baseline; Test type: Superiority; p = 0.7754, Mixed Model for Repeated Measures; Difference in adjusted means = 0.00, 95% CI 2-sided [-0.03 to 0.03], Standard Error of Mean 0.015
Statistical Analysis 4: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; Parietal Lobe: Change from BL was calculated based on mixed-effect model of repeated measure which included the following covariates and stratification factors = Baseline + APOE e4 status + Study + Analysis Visit + Treatment + Treatment*Analysis Visit + Analysis Visit*Baseline; Test type: Superiority; p = 0.9022, Mixed Model for Repeated Measures; Difference in adjusted means = 0.00, 95% CI 2-sided [-0.05 to 0.05], Standard Error of Mean 0.026

19. Secondary Outcome: DBT Period: Percent Change From Baseline to Week 116 in Cerebrospinal Fluid (CSF) Marker of Disease in a Subset of Participants - Total Tau (tTau)
Description: CSF biomarker tTau has been considered as a general marker of neurodegeneration. An elevation in levels of tau, as well as specific pTau species, is thought to be a marker for progressive cellular degeneration in AD.
Time Frame: Baseline, Week 116
Population: CSF mITT Analysis Set included all participants in the ITT analysis set who had at least one valid quantitative CSF measurement. Overall number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in tTau
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 84 | 91
percent change in tTau | 3.2 [-1.74 to 8.37] | -16.6 [-20.40 to -12.54]
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; [analysis description as in outcome 18, analysis 4]; Test type: Superiority; p < .001, ANCOVA

20. Secondary Outcome: DBT Period: Percent Change From Baseline to Week 116 in CSF Marker of Disease in a Subset of Participants - Phosphorylated Tau (pTau-181)
Description: CSF phospho-tau is an indicator of neuronal injury and neurodegeneration. CSF biomarker tTau has been considered as a general marker of neurodegeneration. An elevation in levels of pTau species, is thought to be a marker for progressive cellular degeneration in AD.
Time Frame: Baseline, Week 116
Population: CSF modified ITT analysis set included all participants in the ITT analysis set who had at least one valid quantitative CSF measurement. Overall number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in pTau-181
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 84 | 89
percent change in pTau-181 | 1.1 [-3.76 to 6.20] | -25.2 [-28.65 to -21.49]
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; Test type: Superiority; p < .001, ANCOVA

21. Secondary Outcome: DBT Period: Percent Change From Baseline to Week 116 in CSF Marker of Disease in a Subset of Participants - Neurofilament Light Chain (NFL)
Description: NFL is a neuronal cytoplasmic protein highly expressed in large, myelinated axons. Its levels increase in CSF and blood proportionally to the degree of axonal damage in a variety of neurological disorders, including AD.
Time Frame: Baseline, Week 116
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in NFL
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 85 | 93
percent change in NFL | 15.8 [9.67 to 22.32] | 12.1 [6.41 to 18.11]
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; Test type: Superiority; p = 0.396, ANCOVA

22. Secondary Outcome: DBT Period: Percent Change From Baseline to Week 116 in CSF Marker of Disease in a Subset of Participants - Neurogranin
Time Frame: Baseline, Week 116
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in neurogranin
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab
Number analyzed (Participants) | 84 | 93
percent change in neurogranin | -0.6 [-5.93 to 5.05] | -22.3 [-26.28 to -18.13]
Statistical Analysis 1: Comparison: Global - DBT Period: Placebo vs Global - DBT Period: Gantenerumab; Test type: Superiority; p < .001, ANCOVA

23. Secondary Outcome: China - DBT Period: Change From Baseline to Week 116 in ADAS-Cog13 Score
Description: as for outcome 3
Time Frame: Baseline, Week 116
Population: as for outcome 2
Arm/Group | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: China - DBT Period: Change From Baseline to Week 116 in ADCS-ADL Total Score
Description: ADCS-ADL is a 23-item rater-administered, ObsRO that captures a participant's ability to perform basic activities of daily living (e.g., eating and toileting) and more complex ADL or instrumental activities of daily living (iADL, e.g., using the telephone, managing finances, preparing a meal). Total score ranges from 0-78, with higher scores reflecting better functioning. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 2
Arm/Group | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: China - DBT Period: Change From Baseline to Week 116 in FAQ Score
Description: as for outcome 5
Time Frame: Baseline, Week 116
Population: as for outcome 2
Arm/Group | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: China - DBT Period: DBT Period: Change From Baseline to Week 116 in MMSE Total Score
Description: MMSE is a rater-administered PerfO that includes a set of standardized questions used to evaluate possible cognitive impairment and help stage the severity level of this impairment. The questions target six areas: orientation, registration, attention, short-term recall, language, and constructional praxis/visuospatial abilities. Total score ranges from 0-30, with lower scores indicating greater impairment. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 2
Arm/Group | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: China - DBT Period: Change From Baseline to Week 116 in ADAS-Cog11 Score
Description: The ADAS-Cog11 was designed to measure cognitive symptom change in participants with AD and consisted of 11 tasks. The standard 11 items (and corresponding score range) were: word recall (0-10), commands (0-5), constructional praxis (0-5), naming objects and fingers (0-5), ideational praxis (0-5), orientation (0-8), word recognition (0-12), spoken language ability (0-5), comprehension of spoken language (0-5), word-finding difficulty (0-5), and remembering test instructions (0-5). The test included 7 performance items and 4 clinician-rated items. The ADAS-Cog11 total score was the sum of all 11 individual items, with a total score ranging from 0 (no impairment) to 70 (severe impairment). Higher scores indicated more severe cognitive impairment. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 116
Population: as for outcome 2
Arm/Group | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: China - DBT Period: Change From Baseline to Week 116 in VFT Score
Description: as for outcome 8
Time Frame: Baseline, Week 116
Population: as for outcome 2
Arm/Group | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: China - DBT Period: Change From Baseline to Week 116 in the Coding (DSST) Subtest
Description: as for outcome 9
Time Frame: Baseline, Week 116
Population: as for outcome 2
Arm/Group | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: China - DBT Period: Number of Participants With at Least One AE
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. Total number of participants with at least one event (AEs) have been reported here.
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 124 weeks)
Population: SE analysis set (China) included all participants enrolled in China in the China extension phase who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab
Number analyzed (Participants) | 33 | 35
Participants | 17 | 24

31. Secondary Outcome: China - DBT Period: Number of Participants With Post-baseline Suicidal Ideation or Suicidal Behavior as Measured Using C-SSRS
Description: as for outcome 12
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 124 weeks)
Population: SE analysis set (China) included all participants enrolled in China in the China extension phase who received at least one dose of study drug. Overall number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab
Number analyzed (Participants) | 25 | 30
Participants
  Suicidal Ideation: Passive | 1 | 1
  Suicidal Ideation: Active-Nonspecific (no method, intent, or plan) | 0 | 1
  Suicidal Ideation: Active-Method and intent, but no plan | 1 | 0
  Suicidal Ideation: No Event | 23 | 28
  Suicidal Behavior: No Event | 25 | 30
  Self-injurious Behavior Without Suicidal Intent: No event | 25 | 30

32. Secondary Outcome: China - DBT Period: Number of Participants With at Least One ARIA-E MRI Finding
Description: as for outcome 13
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 124 weeks)
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab
Number analyzed (Participants) | 33 | 35
Participants | 1 | 4

33. Secondary Outcome: China - DBT Period: Number of Participants With at Least One ARIA-H MRI Finding
Description: as for outcome 14
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 124 weeks)
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab
Number analyzed (Participants) | 33 | 35
Participants | 0 | 1

34. Secondary Outcome: China - DBT Period: Number of Participants With Injection-Site Reactions
Description: as for outcome 15
Time Frame: From Day 1 up to 14 weeks after the last dose of blinded study drug (up to 124 weeks)
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab
Number analyzed (Participants) | 33 | 35
Participants | 0 | 0

35. Secondary Outcome: OLE Period: Number of Participants With at Least One AEs
Description: as for outcome 11
Time Frame: From day of first dose in OLE period up to 14 weeks after the last OLE dose (up to 68 weeks)
Population: SE analysis set included all participants randomized during the global phase who received at least one dose of study drug. In the DBT period, 4 participants randomized to placebo arm received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety analysis set, of which one participant entered OLE period.
Measure: Count of Participants; unit: Participants
Arm/Group | Global - OLE Period: Placebo (DBT) to Gantenerumab | Global - OLE Period: Gantenerumab (DBT) to Gantenerumab
Number analyzed (Participants) | 9 | 20
Participants | 8 | 16

36. Secondary Outcome: OLE Period: Number of Participants With Post-baseline Suicidal Ideation or Suicidal Behavior as Measured Using C-SSRS
Description: as for outcome 12
Time Frame: From day of first dose in OLE period up to 14 weeks after the last OLE dose (up to 68 weeks)
Population: SE analysis set included all participants randomized during the global phase who received at least one dose of study drug. In the DBT period, 4 participants randomized to placebo arm received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety analysis set, of which one participant entered OLE period. Overall number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Global - OLE Period: Placebo (DBT) to Gantenerumab | Global - OLE Period: Gantenerumab (DBT) to Gantenerumab
Number analyzed (Participants) | 6 | 19
Participants
  Suicidal Ideation: Active-Method, but no intent or plan | 0 | 1
  Suicidal Ideation: No Event | 6 | 18
  Suicidal Behavior: No Event | 6 | 19
  Self-injurious Behavior Without Suicidal Intent: No event | 6 | 19

37. Secondary Outcome: OLE Period: Number of Participants With at Least One ARIA-H MRI Finding
Description: as for outcome 14
Time Frame: From day of first dose in OLE period up to 14 weeks after the last OLE dose (up to 68 weeks)
Population: SEMRI analysis set included all participants in SE analysis set who had at least one post-baseline safety MRI scan. In DBT period, 4 participants randomized to placebo arm received at least one dose of gantenerumab and were considered in gantenerumab arm for SE analysis set, of which 1 participant entered OLE period.
Measure: Count of Participants; unit: Participants
Arm/Group | Global - OLE Period: Placebo (DBT) to Gantenerumab | Global - OLE Period: Gantenerumab (DBT) to Gantenerumab
Number analyzed (Participants) | 9 | 20
Participants | 1 | 1

38. Secondary Outcome: OLE Period: Number of Participants With at Least One ARIA-E MRI Finding
Description: as for outcome 13
Time Frame: From day of first dose in OLE period up to 14 weeks after the last OLE dose (up to 68 weeks)
Population: SEMRI analysis set included all participants in SE analysis set who had at least one post-baseline safety MRI scan. In DBT period, 4 participants randomized to placebo arm received at least one dose of gantenerumab and were considered in gantenerumab arm for SE analysis set, of which 1 participant entered OLE period. Overall number analyzed is the number of participants with data available for analysis. Overall number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Global - OLE Period: Placebo (DBT) to Gantenerumab | Global - OLE Period: Gantenerumab (DBT) to Gantenerumab
Number analyzed (Participants) | 9 | 20
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: Global: DBT: Day 1 up to 14 weeks post last dose of blinded study drug (up to 131 weeks), OLE: Day 1 of OLE period up to 14 weeks post last OLE dose (up to 68 weeks); China DBT: Day 1 up to 14 weeks post last dose of blinded study drug (up to 124 weeks) All cause mortality: DBT: Day 1 up to the end of study (up to approximately 164 weeks); OLE period: From OLE Day 1 up to the end of the study (up to approximately 86 weeks)
Description: SE analysis set=all participants randomized during global phase who received at least 1 dose of study drug. In the DBT period, 4 participants randomized to placebo arm received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety evaluable set, of which 1 participant entered OLE period. SE analysis set (China)=all participants enrolled in China in China extension phase & received at least 1 dose of study drug.
Arm/Group | Global - DBT Period: Placebo | Global - DBT Period: Gantenerumab | China Extension - DBT Period: Placebo | China Extension - DBT Period: Gantenerumab | Global - OLE Period: Placebo (DBT) to Gantenerumab | Global - OLE Period: Gantenerumab (DBT) to Gantenerumab
All-Cause Mortality (participants affected / at risk) | 11/481 | 3/503 | 0/33 | 0/35 | 1/9 | 0/20
Serious Adverse Events (participants affected / at risk) | 95/481 | 76/503 | 0/33 | 2/35 | 2/9 | 2/20
Other Adverse Events (participants affected / at risk) | 329/481 | 366/503 | 11/33 | 20/35 | 8/9 | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global - DBT Period: Placebo (N=481) | Global - DBT Period: Gantenerumab (N=503) | China Extension - DBT Period: Placebo (N=33) | China Extension - DBT Period: Gantenerumab (N=35) | Global - OLE Period: Placebo (DBT) to Gantenerumab (N=9) | Global - OLE Period: Gantenerumab (DBT) to Gantenerumab (N=20)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paroxysmal atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 9 (9) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis intestinal perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 0 (0) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clonic convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemianopia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural hygroma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIth nerve paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebrobasilar artery dissection (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychomotor retardation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder diverticulum (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global - DBT Period: Placebo (N=481) | Global - DBT Period: Gantenerumab (N=503) | China Extension - DBT Period: Placebo (N=33) | China Extension - DBT Period: Gantenerumab (N=35) | Global - OLE Period: Placebo (DBT) to Gantenerumab (N=9) | Global - OLE Period: Gantenerumab (DBT) to Gantenerumab (N=20)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 26 (29) | 33 (48) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 17 (20) | 26 (43) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 43 (95) | 94 (392) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 12 (14) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 35 (35) | 26 (26) | 3 (3) | 4 (4) | 1 (1) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 5 (5) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 33 (37) | 46 (60) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 6 (6) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 28 (39) | 30 (37) | 0 (0) | 1 (1) | 1 (3) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 13 (18) | 21 (23) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 62 (82) | 60 (94) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 8 (8) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 (36) | 37 (51) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 40 (51) | 43 (49) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (4) | 13 (15) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 4 (5) | 33 (35) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 5 (5) | 102 (161) | 1 (1) | 4 (5) | 3 (4) | 2 (3)
Dizziness (Nervous system disorders) | 41 (49) | 45 (64) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Focal dyscognitive seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 42 (85) | 60 (99) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Somnolence (Nervous system disorders) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 15 (18) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 19 (21) | 19 (21) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depressed mood (Psychiatric disorders) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 22 (22) | 28 (28) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 21 (23) | 25 (26) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder irritation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 19 (19) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 7 (8) | 8 (8) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 13 (13) | 12 (15) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 35 (38) | 41 (54) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 7 (8) | 12 (13) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 5 (5) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 5 (5) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 9 (10) | 13 (13) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 19 (23) | 19 (24) | 2 (2) | 3 (6) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 6 (6) | 9 (9) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT03444870/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT03444870/SAP_001.pdf